CLINICAL TRIAL: NCT03822520
Title: A Randomized, Open-label, Negative and Positive Control, Crossover Clinical Study to Evaluate Effect on QT/QTc Interval After Multiple Dose of Celecoxib in Healthy Adult Volunteers
Brief Title: Clinical Study to Evaluate Effect on QT/QTc Interval After Multiple Dose of Celecoxib
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Samsung Medical Center (Other)
Responsible Party: Principal Investigator, Jung-Ryul Kim, Professor, Samsung Medical Center
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: 2016-11-053
Record Dates: First submitted 2018-11-08; First posted 2019-01-30 (Actual); Last update posted 2019-01-30 (Actual); Status verified 2019-01

CONDITIONS: Qt Interval, Variation in
MeSH Terms: interventions — Celecoxib; Moxifloxacin; Water

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- Celecoxib, Moxifloxacin, Water in order (Experimental): 1. Intervention Celecoxib: Celecoxib 400 mg capsule and water 150ml by mouth, daily for 6days
     Wash-out period (3~6 days)
  2. Intervention Moxifloxacin: Moxifloxacin 400 mg tablet and water 150ml by mouth, once for one day
     Wash-out period (3~6 days)
  3. Intervention Pure water: Water 150ml by mouth without any drug, once for one day
  Interventions: Drug: Celecoxib; Drug: Moxifloxacin; Other: Water
- Celecoxib, Water, Moxifloxacin in order (Experimental): 1. Intervention Celecoxib: Celecoxib 400 mg capsule and water 150ml by mouth, daily for 6days
     Wash-out period (3~6 days)
  2. Intervention Pure water: Water 150ml by mouth without any drug, once for one day
     Wash-out period (3~6 days)
  3. Intervention Moxifloxacin: Moxifloxacin 400 mg tablet and water 150ml by mouth, once for one day
  Interventions: Drug: Celecoxib; Drug: Moxifloxacin; Other: Water
- Moxifloxacin, Water, Celecoxib in order (Experimental): 1. Intervention Moxifloxacin: Moxifloxacin 400 mg tablet and water 150ml by mouth, once for one day
     Wash-out period (3~6 days)
  2. Intervention Pure water: Water 150ml by mouth without any drug, once for one day
     Wash-out period (3~6 days)
  3. Intervention Celecoxib: Celecoxib 400 mg capsule and water 150ml by mouth, daily for 6days
  Interventions: Drug: Celecoxib; Drug: Moxifloxacin; Other: Water
- Water, Moxifloxacin, Celecoxib in order (Experimental): 1. Intervention Pure water: Water 150ml by mouth without any drug, once for one day
     Wash-out period (3~6 days)
  2. Intervention Moxifloxacin: Moxifloxacin 400 mg tablet and water 150ml by mouth, once for one day
     Wash-out period (3~6 days)
  3. Intervention Celecoxib: Celecoxib 400 mg capsule and water 150ml by mouth, daily for 6days
  Interventions: Drug: Celecoxib; Drug: Moxifloxacin; Other: Water

INTERVENTIONS:
Drug: Celecoxib — Celecoxib 400mg capsule
  Other Names: Celebrex
Drug: Moxifloxacin — Moxifloxacin 400mg tablet
  Other Names: Avelox
Other: Water — Pure water 150ml

SUMMARY:
This study is conducted to evaluate effect on QT/QTc Interval after multiple dose of celecoxib among healthy adult volunteers. It is randomized, open-label, negative and postive control, and crossover study. Volunteers will be mainly checked up through ECG to find out changes of QT/QTc interval during the study.

ELIGIBILITY:
Inclusion Criteria:

* Healthy adults between 19-year-old and 40-year-old during the screening day
* BMI between 19 kg/m² and 30 kg/m² during the screening day
* Be able to give an informed consent form after understanding for reasonable explanation of clinical trial's purpose, contents and characteristics of clinical drugs
* Wiling to participate whole clinical trial periods

Exclusion Criteria:

* Person who is able to clinically affect to the study through ECG result during the screening day
* Has critical issue for Torsade de points from heart failure, hypopotassemia, arrhythmia etc., or family history for long QT syndrome, sudden cardiac death.
* Was suffered, or is suffering from like liver, kidney, digestive system, circulatory system, respiratory system, endocrine system(except diabetes), musculoskeletal, neuropsychiatry, or hemato-oncology etc., which is able to effect on clinical study
* Has allergy which is required the treatment or hypersensitive from drugs such as aspirin, anti-biotics, anti-depressants, etc.
* Was administered any drug of other clinical study within 90 days from the randomization day.
* Donated whole blood within 60days or apheresis within 30 days from the randomization day.
* Took any medicine or oriental medicine within 2 weeks, or general pharmaceuticals within 7 days from the randomization day. (For general pharmaceuticals circumstances, PI could decide whether he/she is suitable for the study)
* No intention to take contraceptive which is approved as clinical way, or is planning on giving their sperm or egg during the whole clinical trial.
* Average alcohol consumption per week: >140g
* Average smoking per day: >20
* Average grapefruit juice consumption per day: >4 glasses
* systolic blood pressure <100 mmHg or >150 mmHg, or diastolic pressure <70 mmHg or >100mmHg
* Over 2 times from the maximum reference interval of AST and ALT levels in the blood.
* eGFR by MDRD from creatinine in the blood is less than 30 mL/min.
* doesn't show negative reaction from HIV Test, B hepatitis test, or C hepatitis test
* For woman, doesn't show negative reaction from pregnancy test
* PI decides the person is not suitable to participate the clinical study with other reasons.

Ages: 19 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 28 (Actual)
Dates: Start 2017-06-30 (Actual); Primary Completion 2018-05-25 (Actual); Study Completion 2018-05-25 (Actual)

PRIMARY OUTCOMES:
Change in QTc interval, read manually | -1 hour, -40 minutes, -20 minutes pre-dose at initial administration day and 1 hour, 2 hours, 3 hours, 4 hours, 6 hours, 8 hours, 12 hours, 16 hours, 24 hours post-dose at last administration day
  which is analyzed at the date of initial and final administration of celecoxib, moxifloxacin, water toward healthy volunteers.

SECONDARY OUTCOMES:
Change in QTc , measured automatically | -1 hour, -40 minutes, -20 minutes pre-dose at initial administration day and 1 hour, 2 hours, 3 hours, 4 hours, 6 hours, 8 hours, 12 hours, 16 hours, 24 hours post-dose at last administration day
  which is analyzed at the date of initial and final administration of celecoxib, moxifloxacin, water toward healthy volunteers.
ventricular rate, measured automatically | -1 hour, -40 minutes, -20 minutes pre-dose at initial administration day and 1 hour, 2 hours, 3 hours, 4 hours, 6 hours, 8 hours, 12 hours, 16 hours, 24 hours post-dose at last administration day
  which is analyzed at the date of initial and final administration of celecoxib, moxifloxacin, water toward healthy volunteers.
PR duration, measured automatically | -1 hour, -40 minutes, -20 minutes pre-dose at initial administration day and 1 hour, 2 hours, 3 hours, 4 hours, 6 hours, 8 hours, 12 hours, 16 hours, 24 hours post-dose at last administration day
  which is analyzed at the date of initial and final administration of celecoxib, moxifloxacin, water toward healthy volunteers.
RR duration, measured automatically | -1 hour, -40 minutes, -20 minutes pre-dose at initial administration day and 1 hour, 2 hours, 3 hours, 4 hours, 6 hours, 8 hours, 12 hours, 16 hours, 24 hours post-dose at last administration day
  which is analyzed at the date of initial and final administration of celecoxib, moxifloxacin, water toward healthy volunteers.
QRS duration, measured automatically | -1 hour, -40 minutes, -20 minutes pre-dose at initial administration day and 1 hour, 2 hours, 3 hours, 4 hours, 6 hours, 8 hours, 12 hours, 16 hours, 24 hours post-dose at last administration day
  which is analyzed at the date of initial and final administration of celecoxib, moxifloxacin, water toward healthy volunteers.
Area under the curve within a dosing interval at steady state | 0 hour pre-dose and 1 hour, 2 hours, 3 hours, 4 hours, 6 hours, 8 hours, 12 hours, 16 hours, 24 hours post-dose at final administration day(Day6)
  which is analyzed at the date of final administration of celecoxib
Maximum concentration at steady state | 0 hour pre-dose and 1 hour, 2 hours, 3 hours, 4 hours, 6 hours, 8 hours, 12 hours, 16 hours, 24 hours post-dose at final administration day(Day6)
  which is analyzed at the date of final administration of celecoxib
Time to maximum concentration at steady state | 0 hour pre-dose and 1 hour, 2 hours, 3 hours, 4 hours, 6 hours, 8 hours, 12 hours, 16 hours, 24 hours post-dose at final administration day(Day6)
  which is analyzed at the date of final administration of celecoxib
Minimum concentration at steady state | 0 hour pre-dose and 1 hour, 2 hours, 3 hours, 4 hours, 6 hours, 8 hours, 12 hours, 16 hours, 24 hours post-dose at final administration day(Day6)
  which is analyzed at the date of final administration of celecoxib
Area under the concentration-time curve time zero to the time of the last quantifiable concentration | 0 hour pre-dose and 1 hour, 2 hours, 3 hours, 4 hours, 6 hours, 8 hours, 12 hours, 16 hours, 24 hours post-dose at final administration day(Day1)
  which is analyzed at the date of final administration of moxifloxacin
Maximum concentration | 0 hour pre-dose and 1 hour, 2 hours, 3 hours, 4 hours, 6 hours, 8 hours, 12 hours, 16 hours, 24 hours post-dose at final administration day(Day1)
  which is analyzed at the date of final administration of moxifloxacin
Time to maximum concentration | 0 hour pre-dose and 1 hour, 2 hours, 3 hours, 4 hours, 6 hours, 8 hours, 12 hours, 16 hours, 24 hours post-dose at final administration day(Day1)
  which is analyzed at the date of final administration of moxifloxacin
Half-life | 0 hour pre-dose and 1 hour, 2 hours, 3 hours, 4 hours, 6 hours, 8 hours, 12 hours, 16 hours, 24 hours post-dose at final administration day(Day1)
  which is analyzed at the date of final administration of moxifloxacin
The apparent clearance | 0 hour pre-dose and 1 hour, 2 hours, 3 hours, 4 hours, 6 hours, 8 hours, 12 hours, 16 hours, 24 hours post-dose at final administration day(Day1)
  which is analyzed at the date of final administration of moxifloxacin

CONTACTS AND LOCATIONS:
Overall Officials: JUNGRYUL KIM, MD, PhD, Principal Investigator — Samsung Medical Center
Locations (1):
- Samsung Medical Center, Seoul, South Korea

REFERENCES:
- [Derived] Kim S, Lee H, Ko JW, Kim JR. Effects of Celecoxib on the QTc Interval: A Thorough QT/QTc Study. Clin Ther. 2019 Nov;41(11):2204-2218. doi: 10.1016/j.clinthera.2019.09.004. Epub 2019 Sep 26. PMID 31564512